CLINICAL TRIAL: NCT02811679
Title: A Phase II Study Of Blinatumomab For The Treatment Of Relapsed Or Refractory Indolent Non-Hodgkin Lymphoma
Brief Title: A Study Of Blinatumomab For The Treatment Of Relapsed Or Refractory Indolent Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed early due to slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Jeffrey Barnes, MD PhD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-118
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blinatumomab (Experimental): Blinatumomab will be administered as a continuous IV infusion through a central venous catheter for a 42 day cycle. Blinatumomab will start with a 7 day infusion at 9mcg/d. If no dose limiting toxicity (table 6.1) after 7 days, the dose will be escalated to 28 mcg/d for 7 additional days. If no dose limiting toxicity (table 6.1) after 14 days, blinatumomab will be infused at a target dose of at 112mcg/d for 28 days. Subjects will be restaged after a 6 week treatment free period by PET CT. All subjects without disease progression will receive an additional 4 week cycle starting at the target dose of 112 mcg/d.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab is a bispecific t cell engaging antibody targeting CD19 and CD3 approved for B cell acute lymphoblastic leukemia
  Other Names: Blincyto

SUMMARY:
This research study is studying Blinatumomab as a possible treatment for Indolent Non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. The overall purpose of this study is to determine if blinatumomab is safe and effective for treating adult subjects with relapsed or refractory indolent B cell NHL.

Blinatumomab will be infused causing T cells to recognize the Cancer and work against them. This approach has been FDA approved for acute lymphocytic leukemia but has not yet been approved for lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically determined B cell NHL that is relapsed or primary refractory after initial therapy.

  * Follicular Lymphoma of any grade
  * Marginal zone lymphoma (extranodal, nodal, or splenic). Patients with gastric MALT must have progressed after H. Pylori therapy and radiation. Patients with splenic MZL must have prior splenectomy.
* At least 1 prior line of chemoimmunotherapy if primary refractory or relapsed with in one year. Subjects who respond to initial therapy for greater than one year must have had at least 2 prior lines of therapy including one line with chemoimmunotherapy including an anti-CD20 monoclonal antibody
* Measurable disease that has not been previously irradiated on PET-CT of at least 1.5cm,
* Age ≥18 years.
* ECOG performance status ≤2 ( see Appendix A)
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥750/mcL
  * platelets ≥75,000/mcL
  * total bilirubin < 2.0 x upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal or 5 X ULN
  * if due to lymphoma infiltration
  * creatinine 2.0 X ULN OR
  * creatinine clearance ≥50 mL/min/1.73 m2 for participants with creatinine levels above 2.0 X ULN .
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy within 3 weeks, rituximab or obinutuzumab within 4 weeks, or radioimmunotherapy within 6 weeks prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier. Subjects actively progressing within that window who have recovered from toxicities of prior therapy are also eligible.
* Autologous stem cell transplantation within 12 weeks prior to study entry
* Prior allogeneic transplant
* Therapeutic doses of corticosteroids within 14 days prior to study entry, defined as >20mg/day pf prednisone, or equivalent. Topical and/or inhaled steroids are permitted.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to blinatumomab
* Subjects with known HIV infection
* Pregnant or lactating subjects.
* Chronic infection with hepatitis B or hepatitis C virus
* History of or current relevant CNS pathology such as epilepsy, seizure, paresis,aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome, psychosis
* Prior history of another malignancy (except for non-melanoma skin cancer, in situ cervical or breast cancer, or localized prostate cancer) unless disease free for at least one year and felt at low risk of relapse by treating physician.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or uncontrolled systemic fungal, bacterial, viral, or other infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Barnes, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blinatumomab
Started | 13
Completed | 3
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 6
Not completed — Early study closure due to slow accrual | 3

BASELINE CHARACTERISTICS:
Arm/Group | Blinatumomab
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Count of participants achieving a complete or partial response according to the revised response criteria for malignant lymphoma (2014).
  A complete response is defined as regression of involved nodes to normal size (1.5 cm or less in their greatest transverse diameter for nodes 1.5 cm or greater before therapy). Involved nodes 1.1 - 1.5 cm in their greatest transverse diameter before treatment must have decreased to less than 1 cm in their greatest transverse diameter after treatment, or by more than 75% in the sum of the products of the greatest diameters (SPD). For a complete response, the spleen, if enlarged before therapy on a CT scan, must also have regressed in size and must not be palpable.
  A partial response is defined as 50% or greater decrease in SPD of up to 6 largest dominant masses. There must also be no new sites of disease or increases in the size of the other nodes, liver, or spleen. Splenic/hepatic nodules must regress by at least 50% in SPD.
Time Frame: at completion of treatment (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 13
Participants | 6

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the duration of time from start of treatment to time of documentation of disease progression according to the revised response criteria for malignant lymphoma (2014), death, or loss to follow-up. Progressive disease is defined as appearance of a new PET positive lesion greater than 1.5 cm in any axis, 50% or greater increase in the sum of the products of the greatest diameters (SPD) of more than one node, 50% or greater increase in longest diameter of a previously identified node less than 1 cm in short axis. There must also be a 50% increase from nadir in the SPD of any previous lesions.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 13
months | 4.0 [2.6 to 33.4]

3. Secondary Outcome: Time To Response Rate
Description: Time to response is defined as the duration of time from start of treatment to the achievement of a complete response (CR) or partial response (PR) according to the revised response criteria for malignant lymphoma (2014).
  A CR is defined as regression of involved nodes to normal size (1.5 cm or less in their greatest transverse diameter for nodes 1.5 cm or greater before therapy). Involved nodes 1.1 - 1.5 cm in their greatest transverse diameter before treatment must have decreased to less than 1 cm in this measure after treatment, or by more than 75% in the sum of the products of the greatest diameters (SPD). For a CR, the spleen, if enlarged before therapy on a CT scan, must also have regressed in size and must not be palpable.
  A PR is defined as 50% or greater decrease in SPD of up to 6 largest dominant masses. There must also be no new sites of disease or increases in the size of the other nodes, liver, or spleen. Splenic/hepatic nodules must regress by at least 50% in SPD.
Time Frame: 4 months
Population: The 5 patients who achieved a response were included in the analysis; those who did not achieve a partial response or better were excluded.
Measure: Median (Full Range); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 5
months | 2.8 [2.4 to 3.4]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from response (complete or partial response according to the revised response criteria for malignant lymphoma 2014) to disease progression, death, or loss to follow-up.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 5
months | 30.0 [11.2 to 59.8]

5. Secondary Outcome: Rate Patients Are Discontinued From The Drug Due to Toxicity
Description: Number of patients who discontinued study treatment early due to one or more toxicities.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 13
Participants | 1

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined the duration of time from start of treatment to time of death or loss to follow up.
Time Frame: 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 13
months | NA [NA to NA] — Median could not be estimated due to an insufficient number of events.

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 3/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinatumomab (N=13)
Encephalopathy (Nervous system disorders) | 3 (4)
Neutrophil count decreased (Investigations) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinatumomab (N=13)
Lymphocyte count decreased (Investigations) | 9 (26)
Anemia (Blood and lymphatic system disorders) | 12 (19)
Investigations - Other, specify (Investigations) | 5 (15)
Fatigue (General disorders) | 12 (14)
Fever (General disorders) | 8 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (13)
White blood cell decreased (Investigations) | 5 (13)
Neutrophil count decreased (Investigations) | 4 (12)
Platelet count decreased (Investigations) | 6 (11)
Headache (Nervous system disorders) | 7 (9)
Nausea (Gastrointestinal disorders) | 6 (7)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (6)
Anxiety (Psychiatric disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Alkaline phosphatase increased (Investigations) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4)
Insomnia (Psychiatric disorders) | 4 (4)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Creatinine increased (Investigations) | 2 (3)
Cytokine release syndrome (Immune system disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Infections and infestations - Other, specify (Infections and infestations) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (3)
Tremor (Nervous system disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 2 (2)
Localized edema (General disorders) | 1 (2)
Lymphocyte count increased (Investigations) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study plan was to enroll 28 subjects, but only 13 subjects were enrolled due to slow accrual and early study closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT02811679/Prot_SAP_000.pdf